CLINICAL TRIAL: NCT06774053
Title: Swiss Prospective Cohort of TRAnsgender and Gender Diverse Individuals - the SPECTRA Study
Acronym: SPECTRA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Luzern (Other)
Responsible Party: Principal Investigator, Bettina Winzeler, PD Dr., University Hospital, Basel, Switzerland
Other Study IDs: 2025-00018
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Transgender Individuals; Gender Incongruence
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Cohort of Transgender and Gender Diverse individuals in Switzerland

SUMMARY:
The goal of this observational study is to understand the factors influencing the well-being and health of transgender and gender-diverse (TGD) individuals undergoing gender-affirming therapies in Switzerland. The study population includes TGD individuals aged 16 and older, at various stages of their medical transition, including those who have discontinued or detransitioned.

The main question is:

What are the key factors influencing the well-being and health outcomes of transgender and gender-diverse individuals undergoing gender-affirming therapies?

Researchers will compare health outcomes across different subgroups, such as those at different stages of transition or detransition, to examine the effects of gender-affirming therapies.

Participants will:

Complete electronic questionnaires assessing gender congruence, quality of life, mental health, and other outcomes.

Provide biological samples (e.g., blood, urine, stool, and skin swabs) for laboratory analysis.

Undergo clinical evaluations related to endocrinology, fertility, dermatology, and urology as part of their routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years and above.
* Established diagnosis of gender incongruence
* Indication for gender affirming therapy or ongoing or discontinued gender affirming therapy

Exclusion Criteria:

* Unable to give informed consent
* Missing commitment or ability to study protocol adherence

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for the SPECTRA study will consist of transgender and gender-diverse (TGD) individuals aged 16 and above, diagnosed with gender incongruence, and receiving care at participating Swiss healthcare centers. Recruitment will start at University Hospital Basel and Lucerne Cantonal Hospital and expand to other centers across Switzerland. The study targets individuals at various stages of medical transition, including those initiating, continuing, or discontinuing gender-affirming therapies. Efforts will ensure inclusion of all gender identities to comprehensively address their unique healthcare needs.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2045-01 (Estimated); Study Completion 2045-01 (Estimated)

PRIMARY OUTCOMES:
Gender Congruence as Assessed by Gender Congruence and Life Satisfaction Scale (GCLS) | From enrollment to every routine follow-up assessment at baseline, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, and annually thereafter

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital of Basel, Basel
  - Cantonal Hospital of Lucerne, Lucerne